CLINICAL TRIAL: NCT04309084
Title: A Phase I Study of Human Placental Hematopoietic Stem Cell Derived Natural Killer Cells (CYNK 001) in Multiple Myeloma Patients Following Autologous Stem Cell Transplant in the Front-line Setting.
Brief Title: Natural Killer Cell (CYNK-001) Infusions in Adults With Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYNK-001-MM-002
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma; Neoplasm, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorder; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Antineoplastic Agents; Analgesics, Non-Narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs
Keywords: CYNK-001; Autologous stem cell transplant; Cell therapy; NK cells; Natural killer cells; Multiple Myeloma; Plasma Cell Myeloma; Plasma Cell Neoplasm; Newly Diagnosed Multiple Myeloma; Minimal Residual Disease; MRD
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: The study will utilize a 3+3 open label design, and will enroll up to three dosing cohorts of CYNK-001 given on Day 2 or Days 2, 7, 14 post ASCT. Once MTD has been determined, the Expansion cohort will commence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I (Experimental): Up to three dosing cohorts of CYNK-001 given on Day 2 or Days 2, 7, 14 post ASCT. Once MTD has been determined, the Expansion cohort will commence.
  Interventions: Biological: CYNK-001

INTERVENTIONS:
Biological: CYNK-001 — CYNK-001 is an allogeneic off the shelf cell therapy enriched for CD56+/CD3- NK cells expanded from human placental CD34+ cells.

SUMMARY:
This study will find the maximum tolerated dose (MTD) of CYNK-001 which contain NK cells derived from human placental CD34+ cells and culture-expanded. CYNK-001 cells will be given post Autologous Stem Cell Transplant (ASCT). The safety of this treatment will be evaluated, and researchers will want to learn if NK cells will help in treating Multiple Myeloma.

ELIGIBILITY:
Subject Inclusion Criteria

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject has eligible disease status:

   Newly diagnosed multiple myeloma undergoing or completed induction therapy prior to undergoing first ASCT and presenting MRD positive by NGS after completion of induction therapy.
2. Subject is > 18 and ≤ 75 years of age at the time of signing the informed consent form (ICF).
3. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
4. Subject is willing and able to adhere to the study schedule and other protocol requirements.
5. Performance status of Eastern Cooperative Oncology Group (ECOG) < 2
6. Ability to be off immunosuppressive drugs for at least 3 days prior to the CYNK-001 cell infusion. Steroids at the equivalent of no more than 5 mg prednisone per day are permissible.
7. Subjects must have autologous peripheral blood stem cell graft available in storage for additional transplant in the event of engraftment failure.
8. Female of childbearing potential (FCBP) must not be pregnant and agree to not becoming pregnant for at least 28 days following the CYNK-001. FCBP must agree to use an adequate method of contraception during the treatment period.

   FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
9. Male subjects must agree to use a condom during sexual contact for at least 28 days following the CYNK-001, even if he has undergone a successful vasectomy.

Subject Exclusion Criteria

The presence of any of the following will exclude a subject from enrollment:

1. Subject has plasma cell leukemia.
2. Subject has non-secretory myeloma.
3. Subject has previously undergone allogeneic stem cell transplant.
4. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
5. Subject has any condition including the presence of laboratory abnormalities which places the subject at unacceptable risk if he or she were to participate in the study.
6. Subject has any condition that confounds the ability to interpret data from the study.
7. Subject has a known sensitivity or allergy to lenalidomide which will limit the subject from receiving the mandatory lenalidomide maintenance as part of the study plan.
8. Subject has aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase ≥ 2.5 x the upper limit of normal (ULN) within 7 days prior to melphalan administration. Transient abnormalities should be discussed with the medical monitor.
9. This eligibility criterion removed with Amendment 1
10. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at screening calculated using the Modification of Diet in Renal Disease Study equation. (Levey, 2006)
11. Subject has a bilirubin level > 2 mg/dL (unless subject has known Gilbert's disease) at screening.
12. Subject has had prior treatment with biologic antineoplastic agents less than 7 days before CYNK-001 infusion and at least 5 half-lives since (excludes melphalan). (Exception will be granted for monoclonal antibodies that are known to have long half-lives, in which case a minimum of 2 weeks from last dose will be required). For agents that have known AEs occurring beyond these specified days after administration, this period must be extended beyond the time during which acute AEs are known to occur. Treating physicians are encouraged to discuss cases with the Medical Monitor.
13. Subject is pregnant or breastfeeding.
14. Subject has new or progressive pulmonary infiltrates or pleural effusion large enough to be detected by chest x-ray or computerized tomography (CT) scan within 2 weeks of CYNK-001 infusion.
15. Subject has active autoimmune disease other than controlled connective tissue disorder or those who are not on active therapy.
16. Subject who is human immunodeficiency virus (HIV) positive is excluded due to increased risk of lethal infections when treated with myeloablative chemotherapy.
17. Subject has history of malignancy, other than MM, unless the subject has been free of disease for > 3 years from the date of signing the ICF. Exceptions include the following noninvasive malignancies:

    1. Basal cell carcinoma of the skin
    2. Squamous cell carcinoma of the skin CYNK-001
    3. Carcinoma in situ of the cervix
    4. Carcinoma in situ of the breast
    5. Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
18. Subject has a history of severe asthma and is presently on chronic medications or has a history of other symptomatic pulmonary disease.
19. Untreated chronic infection or treatment of any infection with systemic antibiotics within 2 weeks prior to melphalan.
20. Subject has any other organ dysfunction (Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade 3 or greater) that will interfere with the administration of the therapy according to this protocol.
21. Subject has a resting left ventricular ejection fraction (LVEF) of < 35% obtained by echocardiography or multigated acquisition scan (MUGA).
22. Subject was treated with an investigational product no less than 28 days before CYNK-001 infusion. Subject must no longer be a participant in the previous interventional study at the time of the CYNK-001 infusion. (Subjects who are under survival follow-up or observation associated with a study are permitted, and if treatment information is collected for this period, "Investigational Study" must be used for capturing the study treatment.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  Safety Assessment of Dose-Limiting Toxicity (DLT)
Maximum Tolerated Dose (MTD) or Maximum Planned Dose (MPD) | Up to 28 days
  Safety Assessment of MTD OR MPD
Adverse Events (AE) | Up to 12 months
  Safety Assessment of AE's
Rate of Minimal Residual Disease (MRD) Negativity | Day 90-100
  Efficacy Assessment of MRD

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) Response | Day 90-100
  Efficacy Assessment of MRD
Time to MRD Response | up to 12 months
  Efficacy Assessment of MRD
International Myeloma Working Group (IMWG) response | up to 12 months
  Efficacy Assessment of response
duration of clinical response | up to 12 months
  Efficacy Assessment of response
Progression-free survival | up to 12 months
  Efficacy Assessment of response
time to progression | up to 12 months
  Efficacy Assessment of response
overall survival | up to 12 months
  Efficacy Assessment of response
Quality of life questionnaire | up to 12 months
  Efficacy Assessment of response

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Kilcoyne, MD, Study Director — Celularity Incorporated
Locations (4):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Washington University, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Institute, Buffalo, New York
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915